CLINICAL TRIAL: NCT05957055
Title: LAMAinDiab - Lisdexamphetamine Vs Methylphenidate for Pediatric Patients with ADHD and Type 1 Diabetes - a Randomized Cross-over Clinical Trial
Brief Title: Lisdexamphetamine Vs Methylphenidate for Pediatric Patients with ADHD and Type 1 Diabetes
Acronym: LAMAinDiab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Collaborators: Medical University of Silesia (Other); Medical University of Gdansk (Other); Institute of Medical Sciences of the University of Opole (Unknown); Pediatric Center of the Central Clinical Hospital of the Medical University of Lodz (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LAMA/2021/1; 2022-001906-24 (EudraCT Number); 2021/ABM/02/00006/P/03 (Other Grant/Funding Number: Medical Research Agency); UR/DBL/D/263/2022 (Other: Office for Registration of Medicinal Products, Medical Devices and Biocidal Products)
Record Dates: First submitted 2023-06-30; First posted 2023-07-24 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Attention Deficit Disorder with Hyperactivity; Diabetes Mellitus, Type 1
Keywords: attention deficit disorder with hyperactivity; diabetes mellitus, type 1; methylphenidate; lisdexamfetamine dimesylate; adolescent; child; glycemic variability; randomized cross-over trial; continuous glucose monitoring
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Diabetes Mellitus, Type 1 | interventions — Lisdexamfetamine Dimesylate; Methylphenidate; 5,10-dihydro-5-methylphenazine

STUDY DESIGN:
Intervention Model Description: Interventional, open, randomized (block randomization stratified by center), assessor masked, cross-over
Who Masked: Outcomes Assessor
Masking Description: ADHD symptoms assessment will be performed with teleconsultation with outcomes assessor blinded for patient's allocation. Patients and their parents/legal guardians will be asked to not share the information with the assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylphenidate first, lisdexamfetamine second (Active Comparator): Initial treatment after PT training - methylphenidate (prolonged-release tablet) once-daily with dose optimization for 5-7 weeks and 6 months total therapy then change to lisdexamfetamine once-daily with dose optimization for 5-7 weeks and 6 months total therapy.
  Interventions: Behavioral: parental training in behavior management; Drug: Methylphenidate
- Lisdexamfetamine first, methylphenidate second (Active Comparator): Initial treatment after PT training - lisdexamfetamine once-daily with dose optimization for 5-7 weeks and 6 months total therapy then change to methylphenidate (prolonged-release tablet) once-daily with dose optimization for 5-7 weeks and 6 months total therapy.
  Interventions: Behavioral: parental training in behavior management; Drug: Lisdexamfetamine

INTERVENTIONS:
Behavioral: parental training in behavior management — Parental training in behavior management - online group sessions (4-6 families within group) with trained specialist, 10 once-weekly sessions. To continue to pharmacotherapy, the parents/legal guardians are required to participate in at least 8 out of 10 sessions.
  Other Names: PT training
Drug: Lisdexamfetamine — Once-daily pharmacotherapy with lisdexamfetamine (608137-32-2, SUB32146), administered orally, for a duration of 6 months with initial dose of 30mg and dose optimization for 5-7 weeks (visits after 1st, 3rd and 5th week of therapy to adjust dose, in 20mg steps).
  Other Names: LDX
  Arms: Lisdexamfetamine first, methylphenidate second
Drug: Methylphenidate — Once-daily pharmacotherapy with methylphenidate (prolonged-release tablet, 298-59-9, SUB03254MIG), administered orally, for a duration of 6 months with initial of 18mg dose optimization for 5-7 weeks (visits after 1st, 3rd and 5th week of therapy to adjust dose, in 18mg steps).
  Other Names: MPH
  Arms: Methylphenidate first, lisdexamfetamine second

SUMMARY:
This clinical trial aims to evaluate the safety and effectiveness of an intervention involving parental training in behaviour management and medication in children with both Type 1 Diabetes (T1D) and Attention Deficit Disorder with Hyperactivity (ADHD). ADHD is a neurodevelopmental disorder that affects around 5% of school-age children and adolescents, while T1D is a chronic disease requiring strict management.

After initial parental training provided for parents/legal guardians, the children will be randomized to one of two cross-over groups, and treated with either lisdexamfetamine or methylphenidate first. After dose optimization for first 5-7 weeks, patients will be treated for 6 months total, after which they will be switched to the other drug.

Researchers will then compare the ADHD symptom severity as measured by Conners 3 questionnaire, and compare the frequency of any adverse events associated with the therapy. As secondary outcomes, patient's T1D control and quality of life will be compared between the two drugs.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, cross-over 2nd phase clinical trial in children and adolescents with attention deficit disorder with hyperactivity (ADHD) and type 1 diabetes mellitus (T1D), conducted in four Polish reference pediatric diabetes centers that together provide care for around 25% of Polish pediatric population with T1D.

T1D is a chronic pediatric disorder that requires intensive treatment with subcutaneous insulin, constant monitoring and frequent decision-making from the patient. Its course may be further complicated by comorbidities such as ADHD, which is present in around 5% of general population and reportedly more common in those with T1D. Despite the recognized need for psychiatric screening in children with T1D, ADHD often remains undiagnosed and untreated, resulting in worse therapy adherence and glycemic control, as well increased risk of life-threatening acute diabetes complications.

Each patient will begin the trial starting with the enrollment appointment, followed by a baseline assessment by a diabetologist and a psychological evaluation. After 2-weeks preliminary observation period, the parents/legal guardians of the patient will start a cycle of 10 meetings (one every week, 90 minutes long). Patients will be enrolled in an online once-weekly parental training in behavior management (PT) for ten weeks. The PT will be carried out in small groups (4-6 families per session) and conducted by a qualified and experienced PT therapist and supplemented with homework and educational materials. Qualification for pharmacological treatment will be carried out for those patients who complete the entire PT cycle, defined as the presence of at least 8 out of 10 meetings confirmed by the trainer. This is the designated expert threshold at which an intervention can be considered as carried out correctly. If the parents/legal guardians do not hold the required number of meetings, they will be allowed to make up for the missing classes during the next series of meetings with another group. If the parents/legal guardians do not attend the missing activities during this trial, the child will be excluded from the study.

After completion of PT, each participant will repeat the psychological evaluation to assess the effects of PT intervention alone on ADHD symptoms severity. Those with sustained clinically-significant ADHD symptoms will be qualified for pharmacological intervention. The patient's will be evaluated on diabetologists visit for contraindications to pharmacotherapy, including urine tests (pregnancy and panel test for substance use), ECG with QT segment assessment (to exclude long QT syndrome) and ophthalmological consultation (to exclude glaucoma). Subsequent and final assessment and qualification will be performed by psychiatrist during the nearest online consultation, after which patients will be randomized to pharmacotherapy groups: methylphenidate (MPH, long-release capsule, standard of care) versus lisdexamfetamine (LDX, investigated treatment).

Dose escalation for each drug will be performed over three (up to four) psychiatric consultations during the initial 5-7 weeks. LDX will be started with 30mg once-daily, administered orally, with dose change increment of 20mg every (after 1st, 3rd, 5th and 7th week, to the maximum of 70mg). MPH will be started with 18mg once-daily, administered orally, with dose change incremental of 18mg (after 1st, 3rd, 5th and 7th week, to the maximum of 54mg).

After the maximum tolerated dose is established, patients will continue pharmacotherapy for 6 months. During that time, treatment safety and efficacy will be evaluated twice - after first 3 months by psychological and diabetes care team's evaluation (with small dose adjustments allowed) and after full course (6 months) of therapy. On-demand psychiatric consultations will be allowed. In addition, during both diabetologists visits each participant will donate a dry blood sample for evaluation of the concentration of an allocated drug, and another sample will be self-collected on the day of the final psychological assessment for that arm to ensure that endpoint measurements are not biased by incidental non-adherence. After the last evaluation, participants will return the unused drug to their diabetes care center and will begin a wash-out period. and the treatment will continue for 6 months.

Qualification for the second arm of pharmacotherapy will be based on the same procedures and consultations which will be performed in parallel with the last diabetologists assessment (this means the participant will be on the drug at that time). Final switch and start of the second drug (LDX or MPH) will be based on psychiatrist decision. Its dose adjustment, safety and efficacy monitoring will follow the same procedures over the next 6 months.

The trial primary endpoint (ADHD symptom severity) will be assessed using the Conners 3.0 questionnaire by an investigator blinded to current treatment. Secondary endpoints will include metabolic control assessed with HbA1c and continuous glucose monitoring, and Quality of Life (QoL, measured by PedsQL). Exploratory endpoints will include school attendance, physical activity and sleep parameters (measured with personal wrist activity monitor), change in ADHD symptoms and diabetes control after PT alone, and change in rate of diabetes complications (severe hypoglycemia and diabetic ketoacidosis - rate and associated length of required inpatient treatment).

The primary goal of the trial is to improve ADHD treatment in children with T1D, and assess if treatment efficacy with lisdexamfetamine compared to methylphenidate may lead to both the psychiatric and metabolic benefits. The trial will provide patients with coordinated T1D and ADHD care, access to ADHD medication and PT (MPH is only partially reimbursed in Poland, LDX is unavailable on the Polish market, and PT is not reimbursed in the standard care).

ELIGIBILITY:
Principal inclusion criteria:

* Age 8-16.5 years at study entry;
* T1D diagnosed on the basis of clinical features, presence of autoantibodies typical for type 1 diabetes (at least one of the following: anti-glutamate decarboxylase, islet cell antibody, insulin autoantibody/islet antigen 2 autoantibody, zinc transporter 8 antibody) and/or low C-peptide levels (according to the laboratory standard appropriate for the assay method) and criteria for the diagnosis of diabetes according to the criteria of the Polish Diabetes Association and international societies:

  * an incidental glycemia ≥200mg/dl and symptoms of hyperglycemia (such as increased thirst, polyuria, weakness) or
  * two times a fasting blood glucose ≥125mg/dl or
  * a blood glucose ≥200mg/dL in the 120th minute of an oral glucose load test or
  * HbA1c ≥6.5%.
* T1D diagnosed at least 12 months before recruitment;
* T1D treated with functional intensive insulin therapy
* a diagnosis of ADHD according to Diagnostic and Statistical Manual 5 (DSM-5) criteria confirmed by a psychiatrist or a diagnosis of ADHD according to other criteria recognized in Poland, confirmed by an authorized person as consistent with DSM-5
* Polish citizenship and Polish health insurance

Principal exclusion criteria:

* Daily insulin dose<0.3 j/kg and concomitant HbA1c measurement ≤6.5% from the last 3 months (clinical partial remission of T1D);
* Severely unsatisfactory glycemic control - mean HbA1c over the past year ≥12% (not including HbA1c measurement at diagnosis of T1D);
* Diagnosed intellectual or other disability that prevents participation in the trial or adherence to its therapeutic regimen;
* Clinically apparent cardiovascular disease: recognized hemodynamically significant heart defect, advanced vascular atherosclerosis;
* Diagnosis of other mental illness or disorder preventing participation in the trial, e.g. bipolar affective disorder, schizophrenia, other psychotic disorders, psychoactive substance abuse;
* Diagnosed allergy or hypersensitivity to drugs used in pharmacological intervention -methylphenidate and/or lisdexamphetamine;
* Language barrier making it impossible to conduct a full psychological consultation in Polish;
* Lack of permanent residence in Poland;
* Contraindications as reported for investigated drugs: documented hypertension (at least stage 2), positive family history for sudden cardiac deaths and atrial arrythmias in relatives below 40 y.o., clinically evident glaucoma or abnormally elevated intraocular pressure, history of suicide attempts or present suicide intentions, oppositional defiant disorder, chronic motor tics or Tourette syndrome, pregnancy or breastfeeding, short stature, underweight (≤ 3rd percentile for reference percentile charts), epilepsy, pheochromocytoma, substance abuse or positive drug test results, prolonged treatment with sedative drugs (e.g., 1st generation antihistamines);
* Declared by the parents/legal guardians' inability or unwillingness to come to the Center at the time specified by the protocol, in particular - to pick up the Trial drugs at the dose adjustment stage (the need to pick up 4-5 times over 6-8 weeks, each time within 2-3 days of receiving the recommendations);
* Other reasons that, in the opinion of the attending physician, are more likely to result in difficulties in maintaining the continuity of the participant's participation in the trial or harm to the participant's health in case of participation in the trial.

Ages: 8 Years to 198 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in ADHD symptom scores on the "inattention" scale of the Conners 3 questionnaire | Before pharmacotherapy (after completion of PT training) and the end of the 6-month course of pharmacotherapy with LDX or MPH; similar difference (before pharmacotherapy and after 6 months of therapy) for the other drug
  Change of ADHD symptom severity, measured as the difference in ADHD symptom score on the "inattention" scale of the Conners 3 questionnaire (completed by patient and parent/legal guardian), assessed by the investigator blinded to patient allocation.
Change in ADHD symptom scores on the "hyperactivity/impulsivity" scale of the Conners 3 questionnaire | Before pharmacotherapy (after completion of PT training) and the end of the 6-month course of pharmacotherapy with LDX or MPH; similar difference (before pharmacotherapy and after 6 months of therapy) for the other drug
  Change of ADHD symptom severity, measured as the difference in ADHD symptom score on the "hyperactivity/impulsivity" scale of the Conners 3 questionnaire (completed by patient and parent/legal guardian), assessed by the investigator blinded to patient allocation.
The number of adverse events - methylphenidate arm | Events recorded throughout treatment with MPH for 6 months after randomization or cross-over
  The number of adverse events coded following the MedDRA dictionary.
The frequency of adverse events - methylphenidate arm | Events recorded throughout treatment with MPH for 6 months after randomization or cross-over.
  The frequency of adverse events per patient-month coded following the MedDRA dictionary.
The number of adverse events - lisdexamphetamine arm | Events recorded throughout treatment with LDX for 6 months after randomization or cross-over
  The number of adverse events coded following the MedDRA dictionary.
The frequency of adverse events - lisdexamphetamine arm | Events recorded throughout treatment with LDX for 6 months after randomization or cross-over
  The frequency of adverse events per patient-month coded following the MedDRA dictionary.

SECONDARY OUTCOMES:
Change in Type 1 Diabetes Mellitus metabolic control - glycated haemoglobin | Measured after 6 months of MPH or LDX treatment and compared to the measurement before pharmacotherapy (after PT training, week 10th/22nd depending on PT duration)
  Change of metabolic control of Type 1 Diabetes Mellitus, quantified as the difference in glycated haemoglobin (HbA1c).
Change in Type 1 Diabetes Mellitus metabolic control - CGM-derived percentage percentage time in target range 70-180mg/dL | Measured after 6 months of MPH or LDX treatment (using last 14 days before visit) and compared to the measurement before pharmacotherapy (after PT training, week 10th/22nd depending on PT duration, using data from 14 preceding days)
  Change of metabolic control of Type 1 Diabetes Mellitus, quantified as the difference in the continuous glucose monitoring derived parameters: percentage of time patient's sensor glucose values were in the target range (70-180mg/dl).
Change in Type 1 Diabetes Mellitus metabolic control - CGM-derived percentage percentage time below target range <70mg/dL (hypoglycemia) | MMeasured after 6 months of MPH or LDX treatment (using last 14 days before visit) and compared to the measurement before pharmacotherapy (after PT training, week 10th/22nd depending on PT duration, using data from 14 preceding days)
  Change of metabolic control of Type 1 Diabetes Mellitus, quantified as the difference in the continuous glucose monitoring derived parameters: percentage of time patient's sensor glucose values were in the hypoglycemia range (<70mg/dl).
Change in Type 1 Diabetes Mellitus metabolic control - CGM-derived percentage percentage time below target range <54mg/dL (clinically significant hypoglycemia) | Measured after 6 months of MPH or LDX treatment (using last 14 days before visit) and compared to the measurement before pharmacotherapy (after PT training, week 10th/22nd depending on PT duration, using data from 14 preceding days)
  Change of metabolic control of Type 1 Diabetes Mellitus, quantified as the difference in the continuous glucose monitoring derived parameters: percentage of time patient's sensor glucose values were in the clinically significant hypoglycemia range (<54mg/dl).
Change in Type 1 Diabetes Mellitus metabolic control - CGM-derived percentage percentage time above target range >180mg/dL (hyperglycemia) | Measured after 6 months of MPH or LDX treatment (using last 14 days before visit) and compared to the measurement before pharmacotherapy (after PT training, week 10th/22nd depending on PT duration, using data from 14 preceding days)
  Change of metabolic control of Type 1 Diabetes Mellitus, quantified as the difference in the continuous glucose monitoring derived parameters: percentage of time patient's sensor glucose values were in the hyperglycemia range (>180mg/dl).
Change in Type 1 Diabetes Mellitus metabolic control - CGM-derived percentage percentage time above target range >250mg/dL (significant hyperglycemia) | Measured after 6 months of MPH or LDX treatment (using last 14 days before visit) and compared to the measurement before pharmacotherapy (after PT training, week 10th/22nd depending on PT duration, using data from 14 preceding days)
  Change of metabolic control of Type 1 Diabetes Mellitus, quantified as the difference in the continuous glucose monitoring derived parameters: percentage of time patient's sensor glucose values were in the significant hyperglycemia (>250mg/dl) range.
Change in Type 1 Diabetes Mellitus metabolic control - CGM-derived mean sensor glucose | Measured after 6 months of MPH or LDX treatment (using last 14 days before visit) and compared to the measurement before pharmacotherapy (after PT training, week 10th/22nd depending on PT duration, using data from 14 preceding days)
  Change of metabolic control of Type 1 Diabetes Mellitus, quantified as the difference in the continuous glucose monitoring derived parameters: mean sensor glucose
Change in Type 1 Diabetes Mellitus metabolic control - CGM-derived coefficient of variation | Measured after 6 months of MPH or LDX treatment (using last 14 days before visit) and compared to the measurement before pharmacotherapy (after PT training, week 10th/22nd depending on PT duration, using data from 14 preceding days)
  Change of metabolic control of Type 1 Diabetes Mellitus, quantified as the difference in the continuous glucose monitoring derived parameters: coefficient of variation (calculated as the ratio of the standard deviation to mean sensor glucose, expressed as a percentage).
Improvement of the patient's quality of life (QoL) | Improvement of the patient's quality of life (QoL) measured from baseline (within 2 weeks before PT training), after completion of PT training (week 10th/22nd) and after each 6 months of pharmacotherapy arm
  The outcome will be measured using PedsQL 3.2 questionnaires, completed by patient and parent/legal guardian, assessed by an investigator blinded to patient allocation.
Number of trial participants achieving an improvement in ADHD symptom severity on the basis of Conners 3 "inattention" scale | Measured before pharmacotherapy (after completion of PT training) and the end of the 6-month course of pharmacotherapy with LDX or MPH; similar difference (before pharmacotherapy and after 6 months of therapy) for the other drug
  Number of trial participants achieving an improvement in ADHD symptom severity of at least 1/3 of the baseline value at the end of a given pharmacological intervention, assessed separately on the basis of Conners 3 "inattention" scale. Endpoint assessment by an investigator blinded to patient allocation.
Percentage of trial participants achieving an improvement in ADHD symptom severity on the basis of Conners 3 "inattention" scale | Measured before pharmacotherapy (after completion of PT training) and the end of the 6-month course of pharmacotherapy with LDX or MPH; similar difference (before pharmacotherapy and after 6 months of therapy) for the other drug
  Percentage of trial participants achieving an improvement in ADHD symptom severity of at least 1/3 of the baseline value at the end of a given pharmacological intervention, assessed separately on the basis of Conners 3 "inattention" scale. Endpoint assessment by an investigator blinded to patient allocation.
Number of trial participants achieving an improvement in ADHD symptom severity on the basis of Conners 3 "hyperactivity/impulsivity" scale | Measured before pharmacotherapy (after completion of PT training) and the end of the 6-month course of pharmacotherapy with LDX or MPH; similar difference (before pharmacotherapy and after 6 months of therapy) for the other drug
  Number of trial participants achieving an improvement in ADHD symptom severity of at least 1/3 of the baseline value at the end of a given pharmacological intervention, assessed separately on the basis of Conners 3 "hyperactivity/impulsivity" scale. Endpoint assessment by an investigator blinded to patient allocation.
Percentage of trial participants achieving an improvement in ADHD symptom severity on the basis of Conners 3 "hyperactivity/impulsivity" scale | Measured before pharmacotherapy (after completion of PT training) and the end of the 6-month course of pharmacotherapy with LDX or MPH; similar difference (before pharmacotherapy and after 6 months of therapy) for the other drug
  Percentage of trial participants achieving an improvement in ADHD symptom severity of at least 1/3 of the baseline value at the end of a given pharmacological intervention, assessed separately on the basis of Conners 3 "hyperactivity/impulsivity" scale. Endpoint assessment by an investigator blinded to patient allocation.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Butwicka, A/Prof, Principal Investigator — Department of Biostatistics and Translational Medicine, Medical University of Lodz
Locations (1):
- Pediatric Center of the Central Clinical Hospital of the Medical University of Lodz, Lodz, Łódź Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (with Protected Health Information included) will be provided only in case of serious adverse events and suspected unexpected serious adverse reactions and only to applicable regulators and monitor institutions under appropriate regulations and applicable law.

REFERENCES:
- [Background] Michalak A, Chrzanowski J, Kusmierczyk-Koziel H, Klejman E, Blaziak K, Mianowska B, Szadkowska A, Chobot AP, Jarosz-Chobot P, Mysliwiec M, Makowska I, Kalenik A, Zamarlik M, Wolanczyk T, Fendler W, Butwicka A. Lisdexamphetamine versus methylphenidate for paediatric patients with attention-deficit hyperactivity disorder and type 1 diabetes (LAMAinDiab): protocol for a multicentre, randomised cross-over clinical trial in an outpatient telemedicine-supported setting. BMJ Open. 2023 Dec 12;13(12):e078112. doi: 10.1136/bmjopen-2023-078112. PMID 38086595